CLINICAL TRIAL: NCT05223595
Title: A Phase Ib Study to Investigate the Safety, Tolerability and Preliminary Antitumor Activity of Gentuximab in Combination With Almonertinib in Patients With EGFR Mutation-positive Metastatic Non-Small Cell Lung Cancer
Brief Title: A Study of Gentuximab in Combination With Almonertinib in EGFR Mutation-positive Metastatic NSCLC
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Gensci043-Ib-LC
Record Dates: First submitted 2022-01-04; First posted 2022-02-04 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-01

CONDITIONS: Metastatic Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — aumolertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- dose escalation (Experimental): Gentuximab at a dose of 8 mg/kg or 12 mg/kg based on body weight + Almonertinib at a dose of 110mg for one 28-day cycle
  Interventions: Drug: Gentuximab

INTERVENTIONS:
Drug: Gentuximab — Gentuximab: 8mg/kg or 12mg/kg intravenous (IV) infusion administered on Day 1 and 15 of each cycle; Almonertinib: 110 mg orally once daily.
  Other Names: Almonertinib

SUMMARY:
This is a prospective, multicenter, open label study to investigate the safety and efficacy of Gentuximab plus Almonertinib in metastatic NSCLC patients with EGFR mutation-positive.

ELIGIBILITY:
Inclusion Criteria:

1. The subject can understand the process and methods of the study, complete the study in accordance with the protocol and is willing to sign a written informed consent.
2. Cytologically or histologically confirmed diagnosis of Stage IV NSCLC as defined by the American Joint Committee on Cancer Staging Criteria for Lung Cancer (AJCC 8th edition).
3. Phase Ib dose escalation Cohort: Previous genetic tests confirmed EGFR-sensitive mutations, and received one or two generations of EGFR TKI treatment. After drug resistance, it was confirmed to be positive for EGFR T790M mutation by biopsy or free DNA test.

   •Phase Ib expansion Cohort: Eligible for first-line treatment with erlotinib based on documented evidence of tumor harboring an activating EGFR mutation [exon 19 deletion or exon 21 (L858R) substitution mutation].
4. At least one Measurable lesion.
5. ECOG Performance status (PS) score, 0-1 level.
6. Adequate hematologic function, as defined by: Absolute neutrophil count (ANC) ≥1.5×109/L; hemoglobin concentration ≥90g/L; and platelet count ≥80×109/L.

   * Adequate hepatic function, as defined by: ALT ≤ 2.5 × ULN, AST ≤ 2.5 × ULN, TBIL ≤ 1.5 × ULN (liver metastases patients or Gilbert's Syndrome (unconjugated hyperbilirubinemia) patients ALT ≤ 5 × ULN, AST ≤ 5 × ULN, TBIL ≤ 3 × ULN).
   * Adequate renal function, as defined by: serum creatinine level≤ 1.5 × ULN, or creatinine clearance ≥ 50ml / min.
   * 24-hour urine protein quantitation is <1g（24-hour urine protein quantitative test should be performed when urine protein ≥2+ is found during screening visit）.
7. A life expectancy of ≥12 weeks.
8. Aged between 18 and 75 years
9. Subjects (male and female) who have fertility must agree to use reliable contraceptive methods during the trial and in 3 months after the last administration. Female subjects in childbearing age must be negative for blood pregnancy test prior to enrollment.

Exclusion Criteria:

1. History of other malignancies, excluding full treated non-melanoma skin cancer, in-situ cancer.
2. Brain metastases unless asymptomatic, stable for at least 4 weeks, and not requiring steroids for at least 2 weeks prior to start of study treatment.
3. Subject with positive HCV-Ab, Anti-HIV or TP-Ab, or positive HBS-Ag with copies of HBV DNA > ULN.
4. Interstitial lung disease
5. Evidence of major coagulopathy or other obvious bleeding tendency，which， in the Investigator's opinion, makes it undesirable for the patient to participate in the trial
6. Any of the following major cardiovascular disease： myocardial infarction or received coronary artery bypass graft within 6 months before the start of the study treatment uncontrolled congestive heart failure unstable angina within 6 months before the start of the study treatment any clinically important abnormalities in rhythm （sustained ventricular tachycardia, second degree heart block and third degree heart block）
7. Uncontrolled diabetes
8. Uncontrolled hypertension (blood pressures: systolic≥140 mmHg and/or diastolic ≥90 mmHg)
9. Uncontrolled third space effusion (pleural effusion and pericardial effusion need to be drained or increased rapidly after drained in three days) .
10. Evidence of active tuberculosis
11. Prior treatment with third generation EGFR-TKIs
12. Previously administrated with anti-angiogenic drugs.
13. Has received systematic anti-tumor therapy such as chemotherapy, targeted therapy, immunotherapy, endocrine therapy, etc. within 4 weeks or 5 half-lives of the drug (whichever is shorter) before the first dose of investigational drug.
14. Has received any biologics that targeted the immune system, such as TNF antagonist, anakinra, rituximab, abatacept and tocilizumab, etc. within 4 weeks before the first dose of investigational drug.
15. Has received Chinese medicine with anti-cancer indications or immunomodulatory drugs （including thymosin，interferon，interleukin，except for the use of treatment for leural effusion）within 2 weeks before the first dose of investigational drug.
16. Has received attenuated live vaccine with 12 weeks before the first dose of investigational drug or would receive attenuated live vaccine during the study (except of COVID-19 vaccines).
17. Has received any other investigational drugs within 4 weeks before the first dose of investigational drug
18. Has participated in a clinical study of a non-approved experimental agent within 4 weeks before the first dose of drug.
19. Has undergone major surgery within 4 weeks before screening visit (not including needle biopsy, video-assisted thoracic surgery, mediastinoscopy)，or would undergo planned surgery during the study.

    • Has a nonhealing wound, serious ulcer, or unrecovered bone fracture.
20. Has a known serious allergy reaction to EGFR-TKIs or anti-angiogenic drugs.
21. Have any unresolved toxicities from prior therapy greater than Common Terminology Criteria for Adverse Events V5.0 (CTCAE V5.0) grade 1 before the first dose of investigational drug, with the exception of alopecia.
22. Chest radiotherapy within 4 weeks of the first dose of investigational drug or adverse reactions caused by radiotherapy have not recovered to ≤ CTCAE level 1 (except for alopecia).
23. Female subjects who is pregnant (confirmed by urine or serum pregnancy test) or lactating.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2021-04-02 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicities (DLT) | Up to 4 Weeks
  Number of participants with one or more drug-related adverse events (AEs) defined as DLT in the protocol
AEs or SAEs | Baseline through study completion, about 2 years
  Drug-related adverse events (AEs) or any serious adverse events (SAEs)

SECONDARY OUTCOMES:
Cmax | Cycle 1(day1-day 15)& Cycle 2(day 1-day15) & Cycle 3(day 1) & Cycle 4(day 1) (28 days for every cycle)
  Maximum Concentration
AUC | Cycle 1(day1-day 15)& Cycle 2(day 1-day15) & Cycle 3(day 1) & Cycle 4(day 1) (28 days for every cycle)
  Area Under the Concentration-Time Curve
Objective response rate（ORR） | From date of first dosing until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years
  ORR is defined as the percentage of patients who have at least 1 response of CR or PR prior to any evidence of progression.
Progression-free survival (PFS) | From date of first dosing until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years
  PFS is defined as the time from randomization until the date of objective disease progression or death (by any cause in the absence of progression)
Disease control rate (DCR) | From date of first dosing until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years
  The DCR is defined as the proportion of patients with a best overall response of CR, PR, or SD
Anti-drug antibody number of participants With Anti-drug Antibodies | Cycle 1(day1-day 15)& Cycle 2(day 1) & Cycle 3(day 1) & Cycle 4(day 1) (28 days for every cycle)
  Number of participants with anti-drug antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Shun Lu, Doctor, Principal Investigator — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China